CLINICAL TRIAL: NCT06404593
Title: Dynamic ctDNA Detection for Guiding Adjuvant Therapy and Recurrence Monitoring After Curative Resection of Colorectal Cancer Liver Metastases: A Prospective Study
Brief Title: Dynamic ctDNA Detection for Colorectal Cancer Liver Metastases
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PKUCRLM-1
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Liver Metastases; Colorectal Cancer; Surgery; Circulating Tumor DNA; Minimal Residual Disease
Keywords: Minimal Residual Disease; Colorectal Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm, Residual | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Blood sampling 7 days after surgery
  Interventions: Diagnostic Test: Blood sampling
- Group 2: Blood sampling 1 month after surgery
  Interventions: Diagnostic Test: Blood sampling
- Group 3: Blood sampling 3 to 6 months after surgery
  Interventions: Diagnostic Test: Blood sampling
- Group 4: Blood sampling 6 to 9 months after surgery
  Interventions: Diagnostic Test: Blood sampling
- Group 5: Blood sampling 9 to 12 months after surgery
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Evaluating the value of dynamic monitoring of a colorectal cancer liver metastasis cohort after receiving multipoint ctDNA detecting in predicting recurrence prognosis and guiding adjuvant chemotherapy treatment.

SUMMARY:
Evaluating the value of dynamic monitoring of a colorectal cancer liver metastasis cohort underwent curative resection after receiving multipoint ctDNA detecting in predicting recurrence prognosis and guiding adjuvant chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Before implementing any trial-related procedures, written informed consent should be signed;
2. >=20 and <= 85 years old, male or female;
3. Patients with liver metastases pathologically confirmed as colorectal adenocarcinoma;
4. According to the Response Evaluation Criteria for Solid Tumors (RECIST version 1.1), there is at least one lesion that can be measured by imaging;
5. The multidisciplinary team (MDT) confirmed that the liver metastases were initially resectable ,without locally treatable extrahepatic metastases;
6. The general physical condition is good (ECOG score 0-1);
7. Life expectancy of more than 3 months;
8. There is no obvious symptoms of primary bleeding, obstruction and other indications for emergency surgery;
9. adequate organ function;
10. samples meet NGS quality control requirements;
11. The subjects are able and willing to comply with the visits, treatment plans, laboratory tests and other research-related procedures stipulated in the research protocol.

Exclusion Criteria:

1. Patients who are intolerant to systemic chemotherapy or surgery;
2. Patients with multiple primary lesions;
3. Blood samples and/or baseline tissue samples that do not meet the requirements for testing (hemolysis, low tumor cell content, insufficient DNA extraction yield, etc.);
4. Excessive tissue necrosis after conversion therapy, making it impossible to sample according to testing requirements
5. Patients who have not undergone surgery after conversion therapy, only receiving radiofrequency ablation or chemotherapy follow-up
6. Not all metastatic lesions were resected after conversion therapy, or liver metastatic lesions did not achieve R0 resection
7. No definite mutations detected in the tissue, or mutations detected in tumor tissue were not covered by the designed small panel.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled patients with colorectal liver metastases undergoing radical resection at Hepatopancreatobiliary Surgery Department I of Peking University Cancer Hospital.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 1 year
overall survival | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided